CLINICAL TRIAL: NCT00134654
Title: A Phase II Trial of Two Doses of Conjugated Estrogens (Premarin) in Patients With Androgen-Independent Prostate Cancer
Brief Title: Two Doses of Conjugated Estrogen (Premarin) in Patients With Androgen-Independent Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Beth Israel Deaconess Medical Center (Other); Massachusetts General Hospital (Other); Brigham and Women's Hospital (Other); Lowell General Hospital (Other); South Shore Hospital (Other); Emerson Hospital, Concord, MA (Other); Saint Anne's Hospital (Other)
Responsible Party: Mark Pomerantz, MD, Dana-Farber Cancer Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 02-306
Record Dates: First submitted 2005-08-24; First posted 2005-08-25 (Estimated); Last update posted 2011-06-16 (Estimated); Status verified 2011-06

CONDITIONS: Prostate Cancer
Keywords: Androgen-independent prostate cancer; Premarin; conjugated estrogen
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Estrogens, Conjugated (USP)

ARMS (2):
- Group A (Active Comparator): Premarin once a day
  Interventions: Drug: Premarin
- Group B (Active Comparator): Premarin 3 times a day
  Interventions: Drug: Premarin

INTERVENTIONS:
Drug: Premarin — Group A: 1.25mg once a day Group B: 1.25mg three time a day Group A has been closed and participants have been given the option of enrolling in Group B. Treamtment can continue until disease progression or serious side effects.

SUMMARY:
The purpose of this study is to see if Premarin is useful against androgen-independent prostate cancer and to help understand how drugs such as Premarin may work.

DETAILED DESCRIPTION:
Patients will be randomly assigned to one of two study groups (arm A or Arm B). Arm A will receive 1.25mg of Premarin once daily and arm B will receive 1.25mg of Premarin three times a day. Patients will also receive coumadin daily to help prevent thromboembolic disease.

After reviewing the first 30 patients on Arm A, it was determined that arm A (low dose Premarin) was not effective. Arm A was then closed and patients on Arm A were given the choice to switch to Arm B.

Treatment will continue until there is evidence of disease progression or unacceptable side effects.

Every 4 weeks while receiving Premarin, a physical exam and blood work will be performed. Every 12 weeks a CT scan of the abdomen and pelvis and a bone scan will be performed.

Patients will also be encouraged to undergo standard preventative breast irradiation prior to starting Premarin or up to 4 weeks after starting treatment.

ELIGIBILITY:
Inclusion Criteria:

* Documented histologic evidence of prostate cancer.
* Progressive androgen-independent prostate cancer as defined by the Prostate-Specific Antigen (PSA) Working Group after conventional androgen deprivation and antiandrogen withdrawal.
* PSA > 2ng/ml and serum testosterone of < 50ng/ml
* No history of thromboembolic disease within the prior year
* ECOG performance status of 0-2
* Creatinine < 2 x upper limit of normal
* Bilirubin < 2 x upper limit of normal
* AST < 2 x upper limit of normal

Exclusion Criteria:

* Unstable angina or change in anginal symptoms within the past 6 months.
* Prior therapy with estrogens or PC-SPECS.
* Concurrent megestrol acetate or steroid hormones
* Major surgery or radiation therapy within 4 weeks
* Strontium-89 or samarium-153 therapy within 8 weeks

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2003-03; Primary Completion 2005-07 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
To evaluate the efficacy of two different doses of Premarin in the treatment of patients with androgen-independent prostate cancer

SECONDARY OUTCOMES:
To evaluate the safety of Premarin in this patient population | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Mark Pomerantz, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (3):
- United States (3):
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana-Farber Cancer Insitute, Boston, Massachusetts
  - Massachusetts General Hospital, Boston, Massachusetts